CLINICAL TRIAL: NCT02964702
Title: A Multicenter, Single-arm Study of the Efficacy and Safety of a Thrombectomy Device (T-01) for the Treatment of Acute Cerebral Infarction
Brief Title: Thrombectomy Revascularization of Intracranial Vessel OcclusioN by Originating From Japan (TRON1-Japan)
Acronym: TRON1-Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JIMRO Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJSTO-16-01
Record Dates: First submitted 2016-11-09; First posted 2016-11-16 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

ARMS (1):
- Thrombectomy Device(T-01) (Experimental): Mechanical Thrombectomy with T-01
  Interventions: Device: Thrombectomy Device T-01

INTERVENTIONS:
Device: Thrombectomy Device T-01

SUMMARY:
To evaluate the efficacy and safety of catheter-based thrombectomy for reperfusion by removing a thrombus in a cerebral blood vessel in patients with acute cerebral infarction (within 8 hours after onset), in whom intravenous administration of tissue plasminogen activator (t-PA) is not indicated or reperfusion cannot be achieved by intravenous t-PA administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with neurological disorders caused by blood vessel occlusion associated with acute cerebral infarction
2. Patients who can receive treatment within 8 hours after onset of symptoms of acute cerebral infarction
3. Patients in whom intravenous administration of t-PA is not indicated or reperfusion cannot be achieved by intravenous t-PA administration
4. Patients who have accessible occlusion of the middle cerebral artery (M1 or M2 to 3), basilar artery, vertebral artery, posterior cerebral artery (P1 or P2), anterior cerebral artery (A1 to 2), or intracranial internal carotid artery (pre-procedure TICI score, 0 or 1) as determined by angiography
5. Patients with an NIHSS score of 8 to 30
6. Patients with an mRS score of 0 to 2 before onset
7. Patients aged between 20 and 85 years (at the time of informed consent)
8. Patients who are able to provide written consent (signature) or whose legally acceptable representative (a person with parental authority, spouse, guardian, and an individual legally responsible for his/her custody) can provide written consent (signature)

Exclusion Criteria:

1. Patients who manifest the following:

   * Carotid artery dissection
   * Vasculitis
   * An angulated vessel, making it difficult to guide an investigational device
   * Significant (>50%) stenosis, making it difficult to guide an investigational device
   * Acute intracranial hemorrhage
   * Mass lesion or intracranial tumor
   * Widespread early ischemic changes revealed by CT or MRI
2. Patients who have two or more different major cerebrovascular occlusions requiring treatment
3. Patients with an allergy to contrast agents or who cannot receive them or those who have a serious metal allergy
4. Patients who received heparin within 48 hours and have Partial Thromboplastin Time (PTT)/Activated Partial Thromboplastin Time (APTT) > twice the upper limit of normal
5. Patients with known bleeding tendencies or coagulation deficiency or who have received oral anticoagulants (such as warfarin), and who have (PT-) International Normalized Ratio (INR) >3
6. Patients with platelet count <30,000 /mm3
7. Patients with blood glucose levels <50 mg/dL
8. Patients with uncontrolled hypertension (systolic BP >185 mmHg and diastolic BP >110 mmHg)
9. Patients with expected life expectancy <90 days
10. Female patients who are pregnant or breast feeding
11. Patients who are participating in clinical trials of drugs or medical devices
12. Patients disqualified from participation in the study by the investigator (sub-investigator) due to reasons other than the above

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint of the study is rate of immediate post-procedure reperfusion with the device in 2 pathways/device or 3 pathways/vessel measured using Thrombolysis in Cerebrovascular Infarction (TICI) score of 2a or greater. | immediate post procedure
The primary safety endpoint of the study is mortality within 90 days after the procedure | 90 days

SECONDARY OUTCOMES:
Proportion of subjects with newly diagnosed embolism accompanied by immediate post-procedure embolectomy | immediate post-procedure
Rate of reperfusion not accompanied by symptomatic intracranial hemorrhage within 24 hours after the procedure | 24 hours
Proportion of subjects who have modified Rankin Scale (mRS) score of 2 or greater whose National Institute of Health Stroke Scale (NIHSS) score improved by 10 points or more from baseline at 90 days post-procedure | 90 days
Assessment of mRS scores at 90 days post-procedure | 90 days
Assessment of NIHSS scores at 90 days post-procedure | 90 days
Assessment of Barthel Index (BI) scores at 90 days post-procedure | 90 days
Incidence of intracranial hemorrhage including both symptomatic and asymptomatic within 24 hours after the procedure | 24 hours
Incidence of symptomatic intracranial hemorrhage within 24 hours after the procedure | 24 hours
Incidence of asymptomatic intracranial hemorrhage within 24 hours after the procedure | 24 hours
Incidence of device- or procedure-related serious adverse events within 90 days after the procedure | 90 days
Number of any defect in the investigational device | at the time of inspection before procedure, intraoperative and immediate post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sakai, M.D., D.M. Sc, Principal Investigator — Kobe City Medical Center General Hospital
Locations (13):
- Japan (13):
  - Kurume University Hospital, Kurume, Fukuoka
  - Brain Attack Center Ota Memorial Hospital, Fukuyama, Hiroshima
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Ise Red Cross Hospital, Ise, Mie-ken
  - Kohnan Hospital, Sendai, Miyagi
  - National Cerebral and Cardiovascular Center, Suita, Osaka
  - Gifu University Hospital, Gifu
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Wakayama Medical University Hospital, Wakayama
  - Yamagata City Hospital SAISEIKAN, Yamagata